CLINICAL TRIAL: NCT03571984
Title: A Culturally Adapted Positive Health Programme - Moving on After Breast Cancer Plus- for Breast Cancer Survivors: A Feasibility Randomized Controlled Trial
Brief Title: Moving on After Breast Cancer Plus- for Breast Cancer Survivors
Acronym: MovingonABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC001
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer Female; Depression
Keywords: Breast cancer; depression; Moving on ABC Plus; Pakistan
MeSH Terms: conditions — Depression; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moving on ABC Plus (Experimental): Moving on ABC Plus is combination of two interventions. The culturally adapted CBT and Moving on ABC. CBT will be integrated with The Moving on After Breast Cancer (ABC), which has been developed by Dr Anneela Saleem who suffered from breast cancer. The integrated intervention will consist of 12 sessions (60-90 minutes). The first 8 sessions will be delivered weekly and the last four sessions will be delivered fortnightly
  Interventions: Behavioral: Moving on ABC Plus
- Routine Care (No Intervention): This will consist of routine assessment and management as usually conducted by oncology clinics and general practice. GP's will be informed about the psychiatric diagnosis.

INTERVENTIONS:
Behavioral: Moving on ABC Plus — The intervention has two components. CBT Moving on After Breast Cancer
  Arms: Moving on ABC Plus

SUMMARY:
Breast cancer (BC) ranks second among all the types of cancer and is equally common in developing as well as developed countries. Breast cancer is most common type of cancer worldwide and its diagnosis as well as early treatment is associated with distress. The aim of this study is to explore the feasibility of integrating a 'Moving on After Breast Cancer (ABC)' manual developed by service user (Dr A Saleem) with Cognitive Behavior Therapyfor Pakistani women who are breast cancer (BC) survivors attending primary care and oncology services in Pakistan B) refine the Moving on ABC plus so as to develop a culturally appropriate therapeutic programme to be tested in a future definitive randomized controlled trial.

DETAILED DESCRIPTION:
According to an estimate of World Health Organization (2000) cancer was responsible for 12% of all the deaths from all causes worldwide and rate of cancer is expected to increase 50% by the year 2020. In Pakistan every ninth women has a chance of developing breast cancer, which is highest rate in Asia. The estimated incidence rate of breast cancer in Pakistan is 50/100,000. Despite the high association of distress with breast cancer, data on prevalence of depression in women with breast cancer especially in low income countries is limited .

The proposed project consists of two phases: 1) Phase 1: Integration of the two existing interventions Moving On ABC and the Cognitive Behavior Therapy and the refinement of the integrated intervention. 2) Phase 2: Randomized Control Trial (RCT). Sample size of Phase II will be comprised of 50 patients. Patients will be divided into two groups. One group will receive Group moving on ABC Plus intervention and other group will receive routine care. The total sample size of the effectiveness trial 354.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Breast cancer (stage I to stage IV)
* Has completed primary treatment for breast cancer
* Score of 10 or above on PHQ - 9 or GAD - 7
* Age 18 and above

Exclusion Criteria:

* Already diagnosed with any psychiatric illness
* Already taking psychiatric medicines
* Severe cognitive impairment (not able to give consent to take part in intervention)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 354 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Changes from baseline to 4th and 6th month outcome
  Patient Health Questionnaire-9 (PHQ-9) will be used to diagnose depression.Minimum score of PHQ-9 is 0 and maximum score is 27. This scale categorizes depression in 5 different categories: minimal depression (score range 1-4), Mild depression (5-9), Moderate depression (10-14), Moderately severe depression (15-19), and Sever depression (20-27).

SECONDARY OUTCOMES:
Generalized Anxiety Disorder - 7 | Changes from baseline to 4th and 6th month outcome
  This is a short self-report measure to assess the presence and severity of generalized anxiety.
EuroQol-5D (EQ-5D) | Changes from baseline to 4th and 6th month outcome
  EuroQol-5D (EQ-5D), a 5-itme scale, will be used to assess the quality of life. Lower raw score indicates better quality of life
Multidimensional Scale for Perceived Social Support (MSPSS) | Changes from baseline to 4th and 6th month outcome
  Multidimensional Scale for Perceived Social Support (MSPSS) will be used to assess level of social support. Higher scores indicate higher level of support
Intrusive Thoughts Scale | Changes from baseline to 4th and 6th month outcome
  We will measure Breast Cancer distress with the 7 item subscale of the revised Impact of Event Scale which is reported to be sensitive to change in BC survivors who are receiving a CBT intervention
Rosenberg Self Esteem Scale | Changes from baseline to 4th and 6th month outcome
  This is a ten item Likert scale to measure self-esteem. Higher scores indicate better self esteem.
The Functional Assessment of Cancer Therapy - Breast (FACT-B) | Changes from baseline to 4th and 6th month outcome
  This is one of the most widely used scales to measure health-related quality of life in BC patients. Minimum total score on the scale is "0" and maximum score is 148. Higher score on the scale indicate poor quality of life
Client Satisfaction Questionnaire | This will be administered at 4-month follow up
  This is a well validated self-report measure of client/ patient satisfaction with health services. Minimum total score is "1" and maximum score is "32". Higher score indicate higher level of satisfaction with the services.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, MD, Principal Investigator — PILL
Locations (1):
- Civil Hospital, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American cancer society (2010). The global economic cost of cancer. The American Cancer Society, Inc
- [Background] Husain N, Chaudhry I, Raza-ur-Rehman, Ahmed GR. Self-esteem and obsessive compulsive disorder. J Pak Med Assoc. 2014 Jan;64(1):64-8. PMID 24605716